CLINICAL TRIAL: NCT02383615
Title: A Comparison of Two Different Ultrasound-Guided Approaches to the Saphenous Nerve Block - Adductor Canal vs. Distal Trans-sartorial: A Prospective, Randomized, Blinded, Non-Inferiority Trial
Brief Title: Comparison of Two Different Ultrasound Guided Techniques for Saphenous Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Anil A Marian, Clinical Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201302730
Record Dates: First submitted 2015-02-24; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Efficacy of Ultrasound Guided Nerve Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DTSNB (Active Comparator): Distal transsartorial saphenous nerve block
  Interventions: Procedure: Saphenous nerve block
- ACSNB (Active Comparator): Adductor canal saphenous nerve block
  Interventions: Procedure: Saphenous nerve block

INTERVENTIONS:
Procedure: Saphenous nerve block — Ultrasound guided saphenous nerve blocks with 0.5% Ropivacaine for patients undergoing elective foot and ankle surgery for post-operative pain relief.

SUMMARY:
Saphenous nerve blocks can be technically challenging. Recently described ultrasound techniques have improved the success rate of saphenous nerve blocks, but randomized controlled trials comparing these techniques are lacking. The investigators compared two common ultrasound guided approach for saphenous nerve block: saphenous nerve block at the adductor canal (ACSNB) vs. block by the distal trans-sartorial (DTSNB) approach.

DETAILED DESCRIPTION:
Patients received either ACSNB or DTSNB in this prospective randomized, blinded, non-inferiority clinical trial. The primary objective was to show the non-inferiority of ACSNB to DTSNB in terms of block success. Secondary outcome measures were time required to perform the block, time to onset of successful block, and the visibility of the nerve using ultrasound.

Sample size calculation: To address the primary objective of the study--to show non-inferiority of the ACSNB to DTSNB in terms of success as defined above- the investigators used the test of non-inferiority of two proportions. DTSNB is the primary technique of doing saphenous nerve block at the investigators' institution. From chart review of the electronic records from 2011 to 2012, the investigators found there was a 3% incidence of rescue blocks among saphenous nerve blocks (19 out of 667 blocks) at their institution. This assumed a success rate of approximately 97%. A study by Saranteas et al reported a success rate of 95.6% in healthy volunteers undergoing saphenous nerve block just after it exited from the adductor canal. Based on these two observations, the investigators expected the success rate of DTSNB to be 95%. To establish the non-inferiority of ACSNB to DTSNB, the investigators pre-determined that the success rate of ACSNB should not be lower than 85% (the expected difference in proportions should be less than (95% - 85%) 10%). Under these assumptions, to achieve 80% power, with a one-sided type I error rate of 0.05, the study needed 59 subjects per group; 118 patients total. 120 patients were enrolled for this study., randomized to receive either ACSNB (n=58) or DTSNB (n=62).To show the non-inferiority of the ACSNB to DTSNB, the upper 95% confidence bound of the success rates (πDTSNB - πACSNB) should be less than 10%.

The normality of continuous variables was tested by the Shapiro Wilk's test. Based on the normality assumption, two independent samples t-test or Mann-Whitney U test was performed for continuous variables. Chi-square test or Fisher's exact test was performed for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective foot and ankle surgery receiving saphenous nerve block for pain management
* American Society of Anesthesiologists Physical Status (ASA PS) scores 1, 2 and 3

Exclusion Criteria:

* Neuropathy
* Allergy to local anesthetics
* ASA PS scores 4 and 5

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Success rate of the saphenous nerve block | 30 minutes
  Loss of pin prick sensation to 2 of the 3 pre-defined areas of saphenous nerve distribution in the operative leg after performing the nerve block.

SECONDARY OUTCOMES:
Speed of onset of saphenous nerve block | 30 minutes
  Time taken for loss of pinprick sensation in 2 of the 3 pre-defined areas of saphenous nerve distribution in the leg after performing the nerve block.
Nerve visibility under ultrasound | 30 minutes
  Nerve visibility under ultrasound guidance, graded as 1 (clearly visible) to 3 (not visible even after local anesthetic infiltration)
Time taken to perform block | 30 minutes
  Time taken from skin infiltration of local anesthetic to the nerve block needle removed from patient